CLINICAL TRIAL: NCT05001321
Title: Multi-center and Multi-modal Deep Learning Study of Diagnosis, Therapeutic Outcome and Prognosis of Gastric Cancer
Brief Title: Multi-center and Multi-modal Deep Learning Study of Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: The Second Hospital of Shandong University (Other); Chaoyang Central Hospital (Other); The General Hospital of Fushun Mining Bureau (Unknown); The fourth People's Hospital of Changzhou (Unknown); First Hospital of Jinzhou Medical University (Unknown)
Responsible Party: Principal Investigator, Kai Li, Deputy Director of surgical Oncology, First Hospital of China Medical University
Other Study IDs: FirstHCMU_DL_oncology
Record Dates: First submitted 2021-08-01; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Stomach Neoplasms
Keywords: Diagnosis; Prognosis
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training Group: Based on the inclusion criteria, 2000 gastric cancer patients will be recruited in the analysis. And a model will be constructed based on deep learning.
  Interventions: Radiation: The whole abdomen contrast-enhanced CT scan; Other: H&E stained sections and slides
- Internal Validation Group: Based on the inclusion criteria, 1000 gastric cancer patients will be recruited in this group to verify the sensitivity and specificity of the constructed model.
  Interventions: Radiation: The whole abdomen contrast-enhanced CT scan; Other: H&E stained sections and slides
- External Validation Group: Based on the inclusion criteria, 300 gastric cancer patients from 5 other medical centers will be recruited in this group to verify the sensitivity and specificity of the constructed model.
  Interventions: Radiation: The whole abdomen contrast-enhanced CT scan; Other: H&E stained sections and slides

INTERVENTIONS:
Radiation: The whole abdomen contrast-enhanced CT scan — All the participants were measured by the whole abdomen contrast-enhanced CT scan.
Other: H&E stained sections and slides — HE pathological examination was performed on all specimens of enrolled patients.

SUMMARY:
To assist postoperative pathological diagnosis and classification of gastric cancer by machine learning; To improve the accuracy of pathological diagnosis of gastric cancer by machine learning; To predict the effectiveness of treatment for gastric cancer by deep learning; To construct a model to predict the survival of gastric cancer patients by multimodal deep learning.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of gastric cancer was confirmed by pathology;
* Preoperative enhanced abdominal CT;
* Available detailed clinical and pathological data;
* Integrated follow-up data.

Exclusion Criteria:

* The patients had severe underlying disease;
* Overall survival was less than 3 months;
* No detailed information could be collected.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3000 gastric cancer patients will participate in the phase I study, they will be divided into training group and internal validation group. 300 gastric cancer patients in five other medical centers will form the external validation group.
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum diameter of tumor | 1 day
  To measure the maximum diameter of tumor on preoperative enhanced abdominal CT of patients with gastric cancer.
Growth pattern | 1 day
  To assess the growth pattern on preoperative enhanced abdominal CT of patients with gastric cancer, including endophytic, exophytic and mixed.
Enhancement pattern | 1 day
  To assess the enhancement pattern on preoperative enhanced abdominal CT of patients with gastric cancer, including homogeneous and heterogeneous.
Enhancement degree | 1 day
  To assess the enhancement degree on preoperative enhanced abdominal CT of patients with gastric cancer, including hypoenhancement, isoenhancement and hyperenhancement.
Nucleus size | 1 day
  To obtain the nucleus size of postoperative H&E stained sections and slides of gastric cancer by deep learning.
Nucleus shape | 1 day
  To obtain the nucleus shape of postoperative H&E stained sections and slides of gastric cancer by deep learning.
Distribution of pixel intensity | 1 day
  To obtain the distribution of pixel intensity of postoperative H&E stained sections and slides of gastric cancer by deep learning.
Texture of nuclei | 1 day
  To obtain the texture of nuclei of postoperative H&E stained sections and slides of gastric cancer by deep learning.

SECONDARY OUTCOMES:
Survival status | 1 day
  To analyze the survival status of patients with gastric cancer, involving dead and alive.
Overall survival | 1 day
  To calculate the overall survival of patients with gastric cancer based on days to death and days to last follow-up.
Recurrence/metastasis | 1 day
  To calculate the days to recurrence/metastasis of patients with gastric cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, Principal Investigator — First Hospital of China Medical University
Locations (6):
- China (6):
  - The fourth People's Hospital of Changzhou, Changzhou, Jiangsu
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - The General Hospital of Fushun Mining Bureau, Fushun, Liaoning
  - First Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Second Hospital of Shandong University, Ji'nan, Shandong